CLINICAL TRIAL: NCT00122837
Title: A Comparison of Duloxetine Hydrochloride, Venlafaxine Extended Release, and Placebo in the Treatment of Generalized Anxiety Disorder
Brief Title: A Comparison of Duloxetine Hydrochloride, Marketed Comparator, and Placebo in the Treatment of Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7106; F1J-MC-HMDW
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2007-10-18 (Estimated); Status verified 2007-10

CONDITIONS: Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders | interventions — Duloxetine Hydrochloride; Venlafaxine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine
Drug: venlafaxine
Drug: placebo

SUMMARY:
This is a clinical trial assessing duloxetine and comparator to placebo in patients who have generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients at least 18 years of age, presenting with generalized anxiety disorder (GAD).

Exclusion Criteria:

* Any current and primary Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) Axis I diagnosis other than GAD. Patients diagnosed with major depressive disorder within the past 6 months -or- patients diagnosed with panic disorder, post-traumatic stress disorder, or an eating disorder within the past year -or- obsessive-compulsive disorder, bipolar affective disorder, psychosis factitious disorder, or somatoform disorders during their lifetime
* The presence of an Axis II disorder or history of antisocial behavior, which in the judgement of the investigator would interfere with compliance with study protocol
* Have previously completed or withdrawn from this study or any other study investigating duloxetine or have previously been treated with duloxetine
* History of alcohol or any psychoactive substance abuse or dependence (as defined in the DSM-IV-TR) within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560
Dates: Start 2005-04; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Assess whether duloxetine hydrochloride 60 to 120 mg QD is superior to placebo in the treatment of GAD, defined as statistically greater reduction in anxiety symptoms as measured by the HAMA

SECONDARY OUTCOMES:
Self-reported anxiety symptomatology
Quality of Life
Clinical Global Improvement
HAMA factor scores

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9am-5pm Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Rosario
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Everton Park, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Spring Hill, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Toowoomba, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Armadale, Victoria
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Liège
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Tielt
- Canada (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Toronto, Ontario
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, San Luis Potosí City
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Moscow, Russia
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Taoyuan District
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician. test, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Derived] Perlis RH, Fijal B, Dharia S, Houston JP. Pharmacogenetic investigation of response to duloxetine treatment in generalized anxiety disorder. Pharmacogenomics J. 2013 Jun;13(3):280-5. doi: 10.1038/tpj.2011.62. Epub 2012 Jan 17. PMID 22249355
- [Derived] Sheehan DV, Harnett-Sheehan K, Spann ME, Thompson HF, Prakash A. Assessing remission in major depressive disorder and generalized anxiety disorder clinical trials with the discan metric of the Sheehan disability scale. Int Clin Psychopharmacol. 2011 Mar;26(2):75-83. doi: 10.1097/YIC.0b013e328341bb5f. PMID 21102344
- [Derived] Allgulander C, Nutt D, Detke M, Erickson J, Spann M, Walker D, Ball S, Russell J. A non-inferiority comparison of duloxetine and venlafaxine in the treatment of adult patients with generalized anxiety disorder. J Psychopharmacol. 2008 Jun;22(4):417-25. doi: 10.1177/0269881108091588. PMID 18635722
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com